Metacognitive Training for Negative Symptoms (MCT Minus)

Document date: 2022-12-29

Ethical approval obtained: 2023-04-11

NCT ID: not yet assigned

Author: Dr Linda Swanson, (MA (Hons) Psychology; MSc Clinical Neuropsychology;

Doctorate in Clinical Psychology)

# 1. Purpose and aims

There is a clear rationale for developing interventions targeting negative symptoms of schizophrenia as negative symptoms are a stronger indicator of current and future functioning than positive symptoms (Velligan et al., 2015) and because they respond poorly to medication (Veerman et al., 2017) and existing psychological interventions (Fusar-Poli et al., 2015). This is reflected in the National Institute of Mental Health (NIMH)- Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) consensus statement (Kirkpatrick, Fenton, Carpenter, & Marder, 2006) that emphasised that persistent negative symptoms represent an unmet therapeutic need for patients suffering from schizophrenia.

The purpose of this study is to evaluate, in a scientific manner, the intervention developed by Swanson et al. 2021: Metacognitive Training (MCT) Minus. This intervention adapted MCT to target negative symptoms in psychotic disorders (e.g. schizophrenia, schizoaffective or non-affective functional psychosis) as the original version of MCT (Moritz & Woodward, 2007) focused exclusively on positive symptoms. The specific aim is to study whether MCT Minus is a promising treatment for the intended population in terms of:

- Reductions in negative symptoms as measured by the Clinical Assessment Interview for Negative Symptoms (CAINS) (Forbes et al., 2011), the Motivation and Pleasure Scale- Self-Report (MAP-SR) (Llerena et al., 2013) and the Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1987)
- Reductions in severity of defeatist attitudes as measured by the Dysfunctional Attitudes Scale (DAS) (Weissman & Beck, 1978)
- Improvements in reflective ability as measured by the Reflective Functioning Questionnaire (RFQ-8) (Fonagy et al., 2016)
- Reduction in internalised stigma as measured by the Internalized Stigma of Mental Illness Scale-9 (ISMI-9) (Hammer & Toland, 2017)
- Reductions in depression as measured by the Calgary Depression Scale for Schizophrenia (CDSS) (Addington, Addington, & Schissel, 1990)
- Improved functioning as measured by the World Health Organization (WHO)
  Disability Assessment Schedule (WHODAS) 2.0 (WHO, 2010)

The research will add to existing research by identifying and measuring potential mechanisms of change for negative symptoms (i.e., defeatist attitudes, reflective functioning, stigma and depression). It will also add to the existing evidence base by measuring whether the cognitive biases addressed in MCT lead to changes in the wider conceptualisation of metacognition used elsewhere and whether the promising results seen in the feasibility study of MCT Minus (Swanson et al., 2021) can be replicated in a randomised controlled trial (RCT) with a control group and a blinded assessor. We also hope to replicate the findings of a previous study by Shan et al. 2020, where MCT was found to be related to the modulation of default-mode network (DMN) homogeneity in schizophrenia, an area thought to be involved in self- and other-reflectivity.

### 2. State-of-the-art: Introduction

While clinicians tend to focus on positive symptoms as primary treatment targets in schizophrenia, patients prioritize the treatment of depressive and negative symptoms (Moritz et al., 2017). Persistent negative symptoms are experienced by approximately 20%–40% of individuals diagnosed with schizophrenia (Sarkar et al., 2015). Current research indicates that negative symptoms are independent from positive symptoms, depression, cognitive dysfunctions, and disorganization (Galderisi et al., 2018). However, neither medication nor existing psychosocial interventions have proven to be efficacious in reducing negative symptoms (e.g., Correll & Schooler, 2020; Fusar-Poli et al., 2014; Veerman et al., 2017). Consequently, Lutgens et al. (2017) highlighted the need for better understanding of treatment mechanisms underpinning psychological interventions that directly target negative symptoms.

Psychological conceptualizations suggest that negative symptom expression can, in some cases, be understood as a response to adverse experiences (Aleman et al., 2017). For example, Beck et al.'s (2009) cognitive model suggests that negative symptoms emerge from a process where individuals adopt coping strategies of 'shutting down' the cognitive—affective experience. This allows individuals to cope with overwhelming or aversive situations in the short term but leads to a reliance on negative symptoms (including social withdrawal, avolition, and diminished expression) to reduce exposure to, and impact of, negative experiences in the longer term. From an attachment framework, Griffiths and McLeod (2019) suggest that negative symptoms may be seen 'as responses involving emotional and social withdrawal that emerge from threats to self-security' (p. 62). If negative symptoms can be understood within cognitive and developmental frameworks, it may be possible to develop theoretically driven interventions for their treatment.

### 2.1. A cognitive model of negative symptoms

Negative symptoms are associated with low expectations of future success (Cox et al., 2016), asocial beliefs (Grant & Beck, 2009), a reduced sense of self-efficacy (Bentall et al., 2010), negative self-concepts (Lincoln et al., 2011), defeatist performance beliefs (Campellone et al., 2016) and self-stigma (Horsselenberg et al., 2016). The cognitive model therefore proposes that negative symptoms might be caused and maintained by dysfunctional beliefs arising as a consequence of repeated failures and setbacks. These appraisals might include negative beliefs about social affiliations; low expectations of pleasure, success and acceptance; defeatist beliefs about performance; and a perception of limited resources (see Beck et al., 2019). The self-perception, and perceived self-efficacy, of individuals diagnosed with schizophrenia may also be influenced by self-stigmatizing views of their mental illness. It might be that these factors result in hypervigilance to perceived criticism (Rector et al., 2005). Longitudinal studies have shown support for the cognitive model as defeatist performance attitudes and asocial beliefs are found to predict future negative symptoms (Granholm et al., 2018; Luther et al., 2015; Thomas et al., 2017).

# 2.2. Metacognition and psychosis

Metacognition was initially referred to as the capacity to think about and monitor one's mental processes (Flavell, 1979). However, the definition has broadened in contemporary research (Moritz & Lysaker, 2018), ranging 'from discrete processes involving noticing specific thoughts and feelings to more synthetic acts in which information is integrated into complex representations of the self and others' (García-Mieres et al., 2020, p. 170). This has given rise to interventions targeting metacognitive processes, some of which have been specifically developed for psychosis (e.g., metacognitive training (MCT), Moritz & Woodward, 2007; metacognitive reflection and insight therapy (MERIT), Lysaker & Klion, 2017) while others have been modified for this population (see Lysaker, Gagen, et al., 2020; Moritz et al., 2019;

Weijers et al., 2020). MCT is based on the premise that cognitive biases play a role in the development and maintenance of psychotic symptoms which can be alleviated by targeting underlying cognitive processes (Pos et al., 2018). The aims are to gain insight and to learn practical strategies to manage distressing symptoms (Schneider & Andreou, 2014). MCT has been shown to reduce delusions (Liu et al., 2018) and positive symptoms (Philipp et al., 2019) and improve cognitive insight (Birulés et al., 2020) and biases (Sauvé et al., 2020). Preliminary evidence also suggests effects on quality of life (Moritz, Andreou, et al., 2014) and illness insight (Lopez-Morinigo et al., 2020).

Several authors highlight the links between negative symptoms and compromised capacity for self/others mental state processing (Griffiths & McLeod, 2019; Gumley et al., 2014; Harder, 2014). There is evidence that suggests a link between metacognition and negative symptoms as limitations in complex metacognitive processes predict negative symptoms in first episode psychosis (Austin et al., 2019) and in more chronic samples, even after controlling for defeatist beliefs, affect recognition and neurocognitive functioning (Lysaker et al., 2015). Metacognitive deficits are also associated with concurrent and future negative symptoms when controlling for verbal memory and education (Faith et al., 2020; Lysaker, et al., 2020). Interestingly, self-reflection in itself has been found to mediate the relationship between neurocognition and negative symptoms (especially for deficits in capacity to communicate about internal states, so called diminished expression) while interpersonal cognitive differentiation (i.e., the ability to construe one's experiences as either similar or different from others' experiences) has been found to mediate the pathway between selfreflectivity and negative symptoms (García-Mieres et al., 2019, 2020). This suggests that negative symptom reduction may at least partially depend on improved metacognitive capacity and that a metacognitive intervention specifically targeting negative symptoms may be beneficial.

Swanson et al. (2021) therefore adapted MCT for negative symptoms to assess the acceptability and feasibility of the intervention, examine variable change over the course of the intervention and carry out a preliminary investigation of putative mechanisms of change. The current project is a further evaluation of this, where we hope to achieve similarly encouraging results in a randomised controlled trial (RCT) with a control group and blinding. We also hope to replicate the findings of a previous study by Shan et al. 2020, where MCT was found to be related to the modulation of default-mode network (DMN) homogeneity in schizophrenia, an area thought to be involved in self- and other-reflectivity. Importantly, it was found that high network homogeneity levels at baseline in the bilateral superior medial prefrontal cortex could predict symptomatic improvement after 8 weeks of drug plus psychotherapy treatment; this illustrates that a more developed understanding of the biological mechanisms underlying negative symptoms would allow us to identify patients that would benefit from each type of treatment and, through that, change the prognosis and treatment outcomes of the condition.

# 3. Significance and scientific novelty

Research funding would facilitate a RCT to evaluate the intervention trialled by Swanson et al, 2021 in a more rigorous and scientific manner. Given our limited understanding of negative symptoms and how to treat them (see Galderisi et al., 2021), the study would be of both significance and scientific novelty. To fully understand the biological mechanisms behind negative symptoms is essential to be able to develop future treatment options and to identify patients that would benefit from each type of treatment. A more thorough understanding of schizophrenia would decrease the heterogeneity of the condition which would have vast implications for how individuals diagnosed with schizophrenia are treated both in society and in the healthcare setting.

#### 4. Previous results

Two articles (which were based on the main researcher's doctoral thesis at Edinburgh University with funding from National Health Service (NHS) Lothian) have been published in Clinical Psychology and Psychotherapy (Swanson et al., 2022; Swanson et al. 2022) and a poster has been presented at "The 2022 Congress of the Schizophrenia International, Research Society (SIRS)" (6-10 April 2022 in Florence). The project will also be covered in several articles in "Empati" which is the Schizophrenia Association's paper for members which is also distributed to politicians on local, regional and national level.

## 5. Project description

## 5.1. Participants, sample size, settings and ethics

Eligible participants will be over the age of 18 with a diagnosis of schizophrenia, delusional disorder or non-affective psychosis in Region Sörmland, Region Västmanland and Region Uppland. Exclusion criteria will be evidence of severe organic brain dysfunction or a learning disability, difficulty with the Swedish language, visual and/or hearing impairment, or being unable or unwilling to provide written informed consent. Clinical teams will be approached by L.S. or a research assistant and asked to inform suitable patients about the study. The research assistant will then meet the subjects and inform them (both orally and written) prior to gaining written consent. Subjects who have been allocated to the control group (i.e. supportive counselling) will be offered metacognitive training after the trial has finished if they request this. We have used t/z-test, with a power of 0,85, and a significance level of 0,05, to calculate sample size. In order to find a difference of 4 units on CAINS (as a change in total score of 4 points has been found to show a true change at a 95% confidence level in previous research (Laraki et al., 2022)), 41 participants in each arm will be needed. We will aim to recruit 45 in each arm to allow for drop-out, group heterogeneity and to make future analysis (e.g. on. the effect of medication) possible. Ethical approval will be applied for at the Etikprövningsmyndigheten.

#### 5.2. Intervention

The original MCT intervention was adapted to negative symptoms by incorporating psychoeducation and strategies to target the cognitions suggested by the cognitive model (Beck et al., 2009) to be implicated in the development and/or maintenance of negative symptoms (see Table 1). Although some of the strategies have traditionally been used to target positive symptoms, it is assumed that the same reasoning styles lead to negative symptoms through the dysfunctional cognitions discussed previously (e.g., jumping to conclusions in regard to social rejection and a dysfunctional attribution style reinforcing social withdrawal). Metacognitive training for negative symptoms consists of eight sessions, delivered individually as there is evidence indicating that this approach may lead to stronger effect sizes than delivery in a group format (Liu et al., 2018). The developer of MCT (Professor Steffen Moritz) approved the modification.

#### 5.3. Outcome measures

This study will use a combination of interviews and self-rated questionnaires to assess negative symptoms. The primary outcome measures will be the Clinical Assessment Interview for Negative Symptoms (CAINS) (Forbes et al., 2011), the Motivation and Pleasure Scale—Self-Report (MAP-SR) (Llerena et al., 2013), and the Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1987) (with the PANSS negative factor proposed by Wallwork et al. (2012)). The CAINS was chosen as it has been developed to measure negative symptoms as defined by the NIMH consensus development conference (i.e., blunted affect, alogia, anhedonia, asociality and avolition) (Kumari et al., 2017). (We replaced the Brief

Negative Symptom Scale (BNSS) (Kirkpatrick et al., 2010) with CAINS as the BNSS has not been validated or translated into Swedish).

To identify and measure mechanisms of change, four measures will be used: the Dysfunctional Attitudes Scale (DAS) (Weissman & Beck, 1978) to measure the severity of defeatist attitudes; the Reflective Functioning Questionnaire (RFQ-8) (Fonagy et al., 2016) to assess metacognitive capacity; the Calgary Depression Scale for Schizophrenia (CDSS) (Addington et al., 1990) to measure depression; and the Internalized Stigma of Mental Illness Scale-9 (ISMI-9) (Hammer & Toland, 2017) to measure stigma. Finally, the World Health Organization (WHO) Disability Assessment Schedule (WHODAS) 2.0 (WHO, 2010) will be used as this has been suggested to be a more reliable measure than the Global Assessment of Functioning (GAF) (American Psychiatric Association (APA), 1987) for assessing a person's overall functioning (Gspandl et al., 2018).

#### 5.4. Procedure

Written informed consent, relevant demographic information and baseline measures will be completed before beginning the intervention. The Motivation and Pleasure Scale—Self-Report (MAP-SR) (Llerena et al., 2013) will be used to certify that some level of negative symptoms exist prior to the intervention. The patients will be randomised to either MCT Minus and treatment as usual or supportive counselling combined with treatment as usual using an online calculator. Pre-, post-, and follow-up assessments will be conducted by a research assistant who is blind to group allocation. Exit interviews will be held after completing the intervention where a standardized interview schedule (with open-ended questions) will be applied to minimize variations in questions asked while retaining enough flexibility to assess individual experiences (Patton, 1987). The head of the division psychiatry in the regional health board (Region Sörmland) has approved the study and there are structures (e.g. funding, research time, support from clinicians and managers) that would facilitate recruitment and feasibility.

During the pre and post assessment visits, the patients will also undergo a magnetic resonance imaging (MRI) investigation, including anatomical (T1-weighted) imaging, resting-state functional MRI to assess changes in default mode network connectivity after the active compared to control intervention, and additionally diffusion weighted imaging (DWI) and MR spectroscopy (MRS) to relate the functional connectivity findings to structural connectivity and prefrontal glutamate levels.

### 5.5. Contributors and collaborators

Participants will be recruited by research assistants who the main researcher will train in the intervention. The main researcher (L.S.) will analyse transcripts with thematic analysis (which will then be discussed with other research collaborators), undertake the statistical analysis (potentially with support from a statistician) and write the manuscript (potentially with the assistance of others). Associate Professor Persson will assist with the analysis of the brain scans. Professor Cervenka and Doctor Tyrberg will help with recruitment as they work clinically in Region Uppland and Region Västmanland and together with Professor Moritz, Professor Boden and Associate Professor Persson comment on the final article.

## 6. Data analysis and statistics

#### 6.1. Quantitative data

Repeated measures ANCOVA will be used to evaluate changes at pre, post and follow-up analysis due to the repeated-measure nature of the data whilst regression analysis will be used for identifying and measuring potential mechanisms of change for negative symptoms. Missing data on questionnaires will be replaced with case-mean substitution if fewer than 20% of the items were missing as this has been found to be a robust way of handling data missing on an item level (Fox-Wasylyshyn & El-Masri, 2005).

Preprocessing and analysis of fMRI data will be performed in the conn toolbox in Matlab, preprocessing of DWI and MRS data in FSL and LCModel, respectively, or equivalent software.

### 6.2. Qualitative data

Thematic analysis (Braun & Clarke, 2006) will be used to analyse the qualitative data. The interviews will be transcribed and transcripts will be read multiple times for familiarity with the material and to generate an overview of the responses (Mairs et al., 2011). The recordings will then be analysed with thematic analysis conducted according to a standard format (i.e., exploring the feasibility of the intervention and potential mechanisms of change). Themes will be developed, labelled and reviewed to assure that they are representative of the data set. This analysis will be undertaken by the primary researcher and discussed with other research collaborators.

### 7. International and national collaboration

There is a high level of national collaboration in the project as the main researcher (employed by Region Sörmland) is collaborating with Professor Simon Cervenka, Associate Professor Jonas Persson, and Professor Robert Boden at Region Uppsala/Uppsala University and Dr Tyrberg at Region Västmanland/Uppsala University through this research. There is also a longstanding collaboration with Professor Moritz at University Medical Center Hamburg-Eppendorf Department of Psychiatry and Psychotherapy, Hamburg, Germany.

# 8. Clinical significance and implications of the project

The project is of high importance for individuals with psychosis but also for clinicians as there is a lack of treatment options and knowledge about negative symptoms. This has immense financial implications as schizophrenia, which affects approximately one percent of the population, has been estimated to cost Europe €93,9 billion per year (Marcellusi et al., 2018). The intervention, when it has been fully translated and edited, will be available at the official website for MCT (https://clinical-neuropsychology.de/metacognitive\_training-psychosis/) and hence be available free of charge for clinicians all over the world. The articles will be published with open access agreements.

### 9. References

- Addington, D., Addington, J., & Schissel, B. (1990). A depression rating scale for schizophrenics. *Schizophrenia research*, *3*(4), 247-251.
- Aleman, A., Lincoln, T. M., Bruggeman, R., Melle, I., Arends, J., Arango, C., & Knegtering, H. (2017). Treatment of negative symptoms: Where do we stand, and where do we go? *Schizophrenia Research*, *186*, 55–62.
- American Psychiatric Association (APA). (1987). *Diagnostic and statistical manual of mental disorders (3rd edition, revised) (DSM-III-TR)*. APA.
- Austin, S. F., Lysaker, P. H., Jansen, J. E., Trauelsen, A. M., Nielsen, H. G. L., Pedersen, M. B., ... Simonsen, E. (2019). Metacognitive capacity and negative symptoms in first episode psychosis: Evidence of a prospective relationship over a 3-year follow-up. *Journal of Experimental Psychopathology*, 10(1), 2043808718821572.
- Beck, A. T., Rector, N. A., Stolar, N., & Grant, P. (2009). Schizophrenia. cognitive theory, research and therapy. Guilford Press.
- Beck, A. T., Himelstein, R., & Grant, P. M. (2019). In and out of schizophrenia: Activation and deactivation of the negative and positive schemas. *Schizophrenia Research*, 203, 55–61.
- Bentall, R. P., Simpson, P. W., Lee, D. A., Williams, S., Elves, S., Brabbins, C., & Morrison, A. P. (2010). Motivation and avolition in schizophrenia patients: The role of self-efficacy. *Psychosis*, *2*(1), 12–22.
- Birulés, I., Lopez-Carrilero, R., Cuadras, D., Pousa, E., Barrigton, M. L., Barajas, A., Ochoa, S., Lorente-Rovira, E., González-Higueras, F., Grasa, E., Ruiz-Delgado, I., Cid, J., de Apraiz, A., Montserrat, R., Pélaez, T., Moritz, S., & The Spanish Metacognition Study Group. (2020). Cognitive insight in first-episode psychosis: Changes during metacognitive training. *Journal of Personalized Medicine*, *10*(*4*), 253.
- Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. *Qualitative Research in Psychology*, *3*(2), 77–101.
- Campellone, T. R., Sanchez, A. H., & Kring, A. M. (2016). Defeatist performance beliefs, negative symptoms, and functional outcome in schizophrenia: A meta-analytic review. *Schizophrenia Bulletin*, *42*(6), 1343–1352.
- Cox, C., Jolley, S., & Johns, L. (2016). Understanding and treating amotivation in people with psychosis: An experimental study of the role of guided imagery. *Psychiatry Research*, *246*, 387–391.
- Correll, C. U., & Schooler, N. R. (2020). Negative Symptoms in Schizophrenia: A Review and Clinical Guide for Recognition, Assessment, and Treatment. *Neuropsychiatric Disease and Treatment*, *16*, 519–534.
- Faith, L. A., Lecomte, T., Corbière, M., Francoeur, A., Hache-Labelle, C., & Lysaker, P. H. (2020). Metacognition is uniquely related to concurrent and prospective assessments of negative symptoms independent of verbal memory in serious mental illness. *The Journal of Nervous and Mental Disease*, 208(11), 837–842.
- Flavell, J. H. (1979). Metacognition and cognitive monitoring: A new area of cognitive—developmental inquiry. *American Psychologist*, *34(10)*, 906–911.
- Fonagy, P., Luyten, P., Moulton-Perkins, A., Lee, Y.-W., Warren, F., Howard, S., Ghinai, R., Fearon, P., & Lowyck, B. (2016). Development and validation of a self-report measure of mentalizing: The Reflective Functioning Questionnaire. *PLoS ONE*, 11, e0158678.
- Forbes, C., Blanchard, J. J., Bennett, M., Horan, W. P., Kring, A., & Gur, R. (2010). Initial development and preliminary validation of a new negative symptom measure: the Clinical Assessment Interview for Negative Symptoms (CAINS). *Schizophrenia research*, *124(1-3)*, 36-42.
- Fox-Wasylyshyn, S. M., & El-Masri, M. M. (2005). Handling missing data in self-report measures. *Research in Nursing & Health*, 28(6), 488–495.
- Fusar-Poli, P., Papanastasiou, E., Stahl, D., Rocchetti, M., Carpenter, W., Shergill, S., & McGuire, P. (2014). Treatments of negative symptoms in schizophrenia: meta analysis of 168 randomized placebo-controlled trials. *Schizophrenia Bulletin, 41(4),* 892-899.

- Galderisi, S., Mucci, A., Buchanan, R. W., & Arango, C. (2018). Negative symptoms of schizophrenia: New developments and unanswered research questions. *The Lancet Psychiatry*, *5*(8), 664–677.
- Galderisi, S., Mucci, A., Dollfus, S., Nordentoft, M., Falkai, P., Kaiser, S., ... & Gaebel, W. (2021). EPA guidance on assessment of negative symptoms in schizophrenia. *European Psychiatry*, 64(1).
- García-Mieres, H., Lundin, N. B., Minor, K. S., Dimaggio, G., Popolo, R., Cheli, S., & Lysaker, P. H. (2020). A cognitive model of diminished expression in schizophrenia: The interface of metacognition, cognitive symptoms and language disturbances. *Journal of Psychiatric Research*, *131*, 169–176.
- García-Mieres, H., Niño-Robles, N., Ochoa, S., & Feixas, G. (2019). Exploring identity and personal meanings in psychosis using the repertory grid technique: A systematic review. *Clinical Psychology & Psychotherapy*, *26*(*6*), 717–733.
- Granholm, E., Holden, J., & Worley, M. (2018). Improvement in negative symptoms and functioning in cognitive-behavioral social skills training for schizophrenia: Mediation by defeatist performance attitudes and asocial beliefs. *Schizophrenia Bulletin, 44(3),* 653–661. Grant, P. M., & Beck, A. T. (2009). Defeatist beliefs as a mediator of cognitive impairment, negative symptoms, and functioning in schizophrenia. *Schizophrenia Bulletin, 35(4),* 798–
- Griffiths, H., & McLeod, H. (2019). *Promoting recovery from negative symptoms: An attachment theory perspective.* In K. Berry, S. Bucci, & A. N. Danquah (Eds.), Attachment theory and psychosis: Current perspectives and future directions (pp. 62–83). Routledge/Taylor & Francis Group.
- Gspandl, S., Peirson, RP., Nahhas, RW., Skale, TG., & Lehrer, DS. (2018). Comparing Global Assessment of Functioning (GAF) and World Health Organization Disability Assessment Schedule (WHODAS) 2.0 in schizophrenia. *Psychiatry Res* (259), 251-253. Gumley, A. I., Taylor, H. E. F., Schwannauer, M., & MacBeth, A. (2014). A systematic review of attachment and psychosis: Measurement, construct validity and outcomes. *Acta Psychiatrica Scandinavica*, 129(4), 257–274.
- Hammer, J. H., & Toland, M. D. (2017). Internal structure and reliability of the Internalized Stigma of Mental Illness Scale (ISMI-29) and brief versions (ISMI-10, ISMI-9) among Americans with depression. *Stigma and Health*, *2*, 159-174.
- Harder, S. (2014). Attachment in schizophrenia—Implications for research, prevention, and treatment. *Schizophrenia Bulletin*, *40*(6), 1189–1193.
- Horsselenberg, E. M., van Busschbach, J. T., Aleman, A., & Pijnenborg, G. H. (2016). Self-stigma and its relationship with victimization, psychotic symptoms and self-esteem among people with schizophrenia spectrum disorders. *PLoS ONE*, *11(10)*, e0149763.
- Kay, S. R., Fiszbein, A., & Opfer, L. A. (1987). The positive and negative syndrome scale (PANSS) for schizophrenia. *Schizophrenia bulletin*, *13*(2), 261-276.
- Kirkpatrick, B., Fenton, W. S., Carpenter, W. T., & Marder, S. R. (2006). The NIMH-MATRICS consensus statement on negative symptoms. *Schizophrenia bulletin*, *32*(2), 214-219
- Kirkpatrick, B., Strauss, G. P., Nguyen, L., Fischer, B. A., Daniel, D. G., Cienfuegos, A., & Marder, S. R. (2010). The brief negative symptom scale: psychometric properties. *Schizophrenia bulletin*, *37*(2), 300-305.
- Kumari, S., Malik, M., Florival, C., Manalai, P., & Sonje, S. (2017). An assessment of five (PANSS, SAPS, SANS, NSA-16, CGI-SCH) commonly used symptoms rating scales in schizophrenia and comparison to newer scales (CAINS, BNSS). *Journal of Addiction Research & Therapy*. *8*(3).
- Lincoln, T. M., Mehl, S., Kesting, M. L., & Rief, W. (2011). Negative symptoms and social cognition: Identifying targets for psychological interventions. *Schizophrenia Bulletin*, *37(2)*, 23–32.
- Liu, Y. C., Tang, C. C., Hung, T. T., Tsai, P. C., & Lin, M. F. (2018). The efficacy of metacognitive training for delusions in patients with schizophrenia: A meta-analysis of

- randomized controlled trials informs evidence-based practice. *Worldviews on Evidence-Based Nursing*, 15(2), 130–139.
- Llerena, K., Park, S. G., McCarthy, J. M., Couture, S. M., Bennett, M. E., & Blanchard, J. J. (2013). The Motivation and Pleasure Scale–Self-Report (MAP-SR): Reliability and validity of a self-report measure of negative symptoms. *Comprehensive psychiatry, 54(5), 568-574*. Lopez-Morinigo, J.-D., Ajnakina, O., Martínez, A. S. E., Escobedo-Aedo, P. J., Ruiz-Ruano, V. G., Sánchez-Alonso, S., Mata-Iturralde, L., Muñoz-Lorenzo, L., Ochoa, S., Baca-García, E., & David, A. S. (2020). Can metacognitive interventions improve insight in schizophrenia spectrum disorders? A systematic review and metaanalysis. *Psychological Medicine, 50,* 2289–2301.
- Lutgens, D., Gariepy, G., & Malla, A. (2017). Psychological and psychosocial interventions for negative symptoms in psychosis: Systematic review and meta-analysis. *The British Journal of Psychiatry*, 210(5), 324–332.
- Luther, L., Fukui, S., Firmin, R. L., McGuire, A. B., White, D. A., Minor, K. S., & Salyers, M. P. (2015). Expectancies of success as a predictor of negative symptoms reduction over 18 months in individuals with schizophrenia. *Psychiatry Research*, 229(1–2), 505–510.
- Lysaker, P. H., Chernov, N., Moiseeva, T., Sozinova, M., Dmitryeva, N., Alyoshin, V., Faith, L. A., Karpenko, O., & Kostyuk, G. (2020). Contrasting metacognitive profiles and their association with negative symptoms in groups with schizophrenia, early psychosis and depression in a Russian sample. *Psychiatry Research*, *291*, 113177.
- Lysaker, P. H., Gagen, E., Klion, R., Zalzala, A., Vohs, J., Faith, L. A., Leonhardt, B., Hamm, J., & Hasson-Ohayon, I. (2020). Metacognitive reflection and insight therapy: A recovery-oriented treatment approach for psychosis. *Psychology Research and Behaviour Management*. *13*, 331–341.
- Lysaker, P. H., & Klion, R. E. (2017). Recovery, meaning-making, and severe mental illness: A comprehensive guide to metacognitive reflection and insight therapy. Routledge. Lysaker, P. H., Kukla, M., Dubreucq, J., Gumley, A., McLeod, H., Vohs, J. L., Buck, K. D., Minor, K. S., Luther, L., Leonhardt, B. L., & Belanger, E. A. (2015). Metacognitive deficits predict future levels of negative symptoms in schizophrenia controlling for neurocognition, affect recognition, and self-expectation of goal attainment. Schizophrenia Research, 168(1), 267–272.
- Mairs, H., Lovell, K., Campbell, M., & Keeley, P. (2011). Development and pilot investigation of behavioral activation for negative symptoms. *Behavior Modification*, *35(5)*, 486–506. Marcellusi, A., Fabiano, G., Viti, R., Morel, P. C. F., Nicolò, G., Siracusano, A., & Mennini, F. S. (2018). Economic burden of schizophrenia in Italy: a probabilistic cost of illness analysis. *BMJ open*, *8(2)*, e018359.
- Moritz, S., Andreou, C., Schneider, B. C., Wittekind, C. E., Menon, M., Balzan, R. P., & Woodward, T. S. (2014). Sowing the seeds of doubt: A narrative review on metacognitive training in schizophrenia. *Clinical Psychology Review, 34(4),* 358–366.
- Moritz, S., Berna, F., Jaeger, S., Westermann, S., & Nagel, M. (2017). The customer is always right? Subjective target symptoms and treatment preferences in patients with psychosis. *European Archives of Psychiatry and Clinical Neuroscience*, 267(4), 335–339.
- Moritz, S., Klein, J. P., Lysaker, P. H., & Mehl, S. (2019). Metacognitive and cognitive-behavioral interventions for psychosis: New developments. *Dialogues in Clinical Neuroscience*, *21*(*3*), 309–317.
- Moritz, S., & Lysaker, P. H. (2018). Metacognition—What did James H. Flavell really say and the implications for the conceptualization and design of metacognitive interventions. *Schizophrenia Research*, *201*, 20–26.
- Moritz, S., & Woodward, T. S. (2007). Metacognitive training for schizophrenia patients (MCT): a pilot study on feasibility, treatment adherence, and subjective efficacy. *German Journal of Psychiatry*, *10*(3), 69-78.
- Patton, M. Q. (1987). How to use qualitative methods in evaluation (Vol. No. 4). Sage. Philipp, R., Kriston, L., Lanio, J., Kühne, F., Härter, M., Moritz, S., & Meister, R. (2019). Effectiveness of metacognitive interventions for mental disorders in adults—A systematic

- review and meta-analysis (METACOG). *Clinical Psychology & Psychotherapy*, 26(2), 227–240.
- Pos, K., Meijer, C. J., Verkerk, O., Ackema, O., Krabbendam, L., & de Haan, L. (2018). Metacognitive training in patients recovering from a first psychosis: An experience sampling study testing treatment effects. *European Archives of Psychiatry and Clinical Neuroscience*, 268(1), 57–64.
- Rector, N. A., Beck, A. T., & Stolar, N. (2005). The negative symptoms of schizophrenia: A cognitive perspective. *The Canadian Journal of Psychiatry*, *50*(*5*), 247–257.
- Sarkar, S., Hillner, K., & Velligan, D. I. (2015). Conceptualization and treatment of negative symptoms in schizophrenia. *World Journal of Psychiatry*, *5*(4), 352–361.
- Sauvé, G., Lavigne, K. M., Pochiet, G., Brodeur, M. B., & Lepage, M. (2020). Efficacy of psychological interventions targeting cognitive biases in schizophrenia: A systematic review and meta-analysis. *Clinical Psychology Review*, 101854.
- Schneider, B. C., & Andreou, C. (2014). A critical review of metacognitive training (MCT) for psychosis: Efficacy, proposed mechanisms of action and significance for functional outcomes. *OA Behavioral Medicine*, 1.
- Strauss, G. P., Keller, W. R., Buchanan, R. W., Gold, J. M., Fischer, B. A., McMahon, R. P., Catalano, L. T., Culbreth, A. J., Carpenter, W. T., & Kirkpatrick, B. (2012). Next-generation negative symptom assessment for clinical trials: Validation of the Brief Negative Symptom Scale. *Schizophrenia Research*, 142(1–3), 88–92.
- Swanson, L., Schwannauer, M., Bird, T., Eliasson, E., Millar, A., Moritz, S., & Griffiths, H. (2021). Metacognitive training modified for negative symptoms: A feasibility study. *Clinical Psychology & Psychotherapy*.
- Thomas, E. C., Luther, L., Zullo, L., Beck, A. T., & Grant, P. M. (2017). From neurocognition to community participation in serious mental illness: The intermediary role of dysfunctional attitudes and motivation. *Psychological Medicine*, *47*(5), 822–836.
- Üstün, T. B., Kostanjsek, N., Chatterji, S., & Rehm, J. (Eds.). (2010). *Measuring health and disability: Manual for WHO disability assessment schedule WHODAS 2.0*. World Health Organization.
- Veerman, S. R., Schulte, P. F., & de Haan, L. (2017). Treatment for Negative Symptoms in Schizophrenia: A Comprehensive Review. *Drugs*, 77(13), 1423-1459.
- Velligan, D. I., Roberts, D., Mintz, J., Maples, N., Li, X., Medellin, E., & Brown, M. (2015). A randomized pilot study of MOtiVation and Enhancement (MOVE) Training for negative symptoms in schizophrenia. *Schizophrenia research*, *165*(2), 175-180.
- Wallwork, R. S., Fortgang, R., Hashimoto, R., Weinberger, D. R., & Dickinson, D. (2012). Searching for a consensus five-factor model of the Positive and Negative Syndrome Scale for schizophrenia. *Schizophrenia Research*, *137(1)*, 246–250.
- Weijers, J. G., Ten Kate, C., Debbané, M., Bateman, A. W., De Jong, S., Selten, J. P., & Eurelings-Bontekoe, E. H. M. (2020). Mentalization and psychosis: A rationale for the use of mentalization theory to understand and treat non-affective psychotic disorder. *Journal of Contemporary Psychotherapy, 50,* 1–10.
- Weissman, A.; Beck, AT. *Development and validation of the Dysfunctional Attitude Scale: A preliminary Investigation*. Paper presented at the Education Research Association; Toronto, Ontario, Canada. 1978.